CLINICAL TRIAL: NCT05683457
Title: A Phase 2, Observer-Blind, Placebo-Controlled Proof-of-Concept Trial to Evaluate Efficacy, Safety, and Immunogenicity of mRNA-1647 Cytomegalovirus Vaccine in Patients Who Have Undergone Allogeneic Hematopoietic Cell Transplantation (HCT)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of mRNA-1647 Cytomegalovirus (CMV) Vaccine in Allogenic Hematopoietic Cell Transplantation (HCT) Participants.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1647-P205
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cytomegalovirus Infection
Keywords: Human cytomegalovirus; Human Herpesvirus; mRNA-1647; Moderna; CMV; Cytomegalovirus Vaccine; Cytomegalovirus Infections; Cytomegalovirus Congenital; Virus Disease; Infection Viral; DNA Virus Infections; Messenger RNA; Hematopoietic cell transplantation
MeSH Terms: conditions — Cytomegalovirus Infections; Herpes Simplex; Virus Diseases; DNA Virus Infections | interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1647 (Experimental): Participants will receive mRNA-1647 by intramuscular (IM) injection on Day 42, Day 67, and Day 92, and a booster dose on Day 180.
  Interventions: Biological: mRNA-1647
- Placebo (Placebo Comparator): Participants will receive mRNA-1647 matching placebo by IM injection on Day 42, Day 67, and Day 92, and a booster dose on Day 180.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1647 — Lyophilized product that is reconstituted with 0.9% sodium chloride (normal saline).
  Arms: mRNA-1647
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The main purpose of the study is to evaluate the efficacy and safety of mRNA-1647 compared to placebo to prevent first clinically significant cytomegalovirus infection (CS-CMVi) in the period following cessation of CMV prophylactic treatment (for example, letermovir) on Day 100 post-HCT through Month 9 post-HCT.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of an allogeneic HCT.
* CMV-seropositive, defined as a documented positive test for anti-CMV IgG.
* High-risk for CMV: HCT from related, unrelated, or haploidentical donor with post-transplant cyclophosphamide for graft-versus-host-disease (GVHD) prophylaxis; or HCT from related or unrelated donor with at least one mismatch at any of the following human leukocyte antigen (HLA) gene loci (HLA-A, B, C, and DRB1); or HCT from related or unrelated donor with myeloablative conditioning.
* Persons of nonchildbearing potential or of childbearing potential with negative urine or serum pregnancy test on the day of first study injection.
* Persons of childbearing potential who have practiced adequate contraception or have abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose.
* Persons of childbearing potential who have agreed to continue adequate contraception or abstain from all activities that could result in pregnancy through 3 months after last study injection.
* Persons who are not currently breast/chestfeeding.
* Willingness to comply with study procedures and provide written informed consent.

Exclusion Criteria:

* History of a diagnosis or condition that, in the judgment of the Investigator, may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* A documented positive human immunodeficiency virus (HIV) test.
* Treatment with alemtuzumab (Campath®), antithymocyte globulin (ATG), or any equivalent in-vivo T cell depleting agent within 12 months.
* HCT with ex-vivo T cell depletion.
* Low risk for CMV: HCT from related or unrelated donor with reduced intensity conditioning (RIC) and no other high-risk features.
* History of prior hematopoietic cell transplantation within 12 months.
* Receipt of prior investigational CMV vaccines or participation in another CMV therapeutic study that may interfere with study outcome measures as determined by the Investigator.
* Suspected or known allergic reaction to any component of any mRNA vaccine or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to the First Occurrence of an CS-CMVi Event as Measured by initiation of anti-CMV Antiviral Therapy | Day 100 to Month 9
Number of Participants with Solicited Local and Systemic Reactogenicity Adverse Reactions (ARs) | Up to Day 187 (7 days after last study injection)
Number of Unsolicited Adverse Events (AEs) | Up to Day 205 (25 days after last study injection)
Number of Participants with Severe AEs | Up to Day 365
Number of Participants with Serious Adverse Events (SAEs) | Up to Day 365
Number of Participants with Grade ≥3 Acute Graft-Versus-Host Disease (GVHD) | Up to Day 365

SECONDARY OUTCOMES:
Number of Participants with First Occurrence of All CS-CMVi Events as Measured by Initiation of Anti-CMV Antiviral and/or End-Organ Disease | Day 100 to Month 9
Number of Participants with an Occurrence of CMV Viremia | Day 100 to Month 9
  CMV Viremia is defined as ≥300 international units/milliliters (IU/mL).
Number of Participants with CMV End-Organ Disease | Day 100 to Month 9
Duration of CMV Viremia | Day 100 to Month 9
Duration of CMV Treatment | Day 100 to Month 9
Number of Participants with Non-Relapse Mortality at 9 Months Post-HCT. | Month 9
Titer of CMV-Specific Neutralizing Antibody (nAb) | Days 42, 67, 92, 117, 180, 205 and 270
Geometric Mean Titer (GMT) of Anti-gB-Specific Immunoglobulin G (IgG) and Anti-Pentamer-Specific IgG as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Days 42, 67, 92, 117, 180, 205 and 270
Geometric Mean Concentration (GMC) of Anti-gB-Specific Immunoglobulin G (IgG) and Anti-Pentamer-Specific IgG as Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | Days 42, 67, 92, 117, 180, 205 and 270
Geometric Mean Fold Rise (GMFR) of Postbaseline/Baseline GMTs or GMCs | Days 42, 67, 92, 117, 180, 205 and 270

CONTACTS AND LOCATIONS:
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States